CLINICAL TRIAL: NCT06516809
Title: The Accuracy of the Dormotech VLAB During Stable Hypoxia Plateaus
Status: Completed | Type: Observational
Sponsor: Dormotech Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: VLAB_SpO2_C_T_1
Record Dates: First submitted 2024-07-15; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: forehead; reflectance; SpO2 sensor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: DormoTech Vlab SpO2 sensor — The Dormotech Vlab sensor was applied to one of the subject's forehead. Reference pulse oximeters were applied to the right fingers. Blood gas analysis to determine hemoglobin saturation (SaO2) was performed using an ABL-90 Flex Plus multi-wavelength oximeter (Hemoximeter, Radiometer, Copenhagen). The ABL90 Flex Plus contains factory calibration standards and automatically performs regular quality controls.

SUMMARY:
The purpose of the study is to determine the accuracy of the Dormotech VLAB (SpO2) Sensor in accordance with the FDA Guidance on Pulse Oximeters - Premarket Notification Submissions [510(k)s], in range of arterial HbO2 saturations from 100% down to 70%.

This was a prospective study with healthy volunteers.

The primary objective of the study was to determine the accuracy of the Dormotech VLAB sensor from saturations from 100 down to 70%. As the primary endpoint, the accuracy of the device during non-motion tests was determined by comparing the pulse oximeter reading during brief, steady-state hypoxia plateaus with a gold-standard measurement of blood oxyhemoglobin saturation (arterial blood sample processed in a multi-wavelength hemoximeter).

DETAILED DESCRIPTION:
The purpose of the study is to determine the accuracy of the Dormotech VLAB (SpO2) Sensor in accordance with the FDA Guidance on Pulse Oximeters - Premarket Notification Submissions [510(k)s], in the range of arterial HbO2 saturations from 100% down to 70%.

The subjects represent a diverse group in terms of age, height, weight, ethnicity, and skin types, which is beneficial for generalizing findings across different demographics. Subjects span all six types, indicating a wide range of skin types from very fair (Type I) to deeply pigmented dark (Type VI).

This was a prospective study with healthy volunteers.

The primary objective of the study was to determine the accuracy of the Dormotech VLAB sensor from saturations from 100 down to 70%. As the primary endpoint, the accuracy of the device during non-motion tests was determined by comparing the pulse oximeter reading during brief, steady-state hypoxia plateaus with a gold-standard measurement of blood oxyhemoglobin saturation (arterial blood sample processed in a multi-wavelength hemoximeter).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or Subject is male or female, aged 18 and < 50.
* Subject is in good health with no evidence of any medical problems.
* Subject is fluent in both written and spoken English.
* Subject has provided informed consent and is willing to comply with the study procedure

Exclusion Criteria:

* Subject is obese (BMI >35).
* Subject has known history of heart disease, lung disease, kidney or liver disease.
* Diagnosis of asthma, sleep apnea, or use of CPAP.
* Subject has diabetes.
* Subject has a clotting disorder.
* Subject uses any anticoagulative medication (blood thinner).
* Subject has a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
* Subject has any other serious systemic illness.
* Subject is a current smoker.
* Subject with any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators would interfere with the sensors working correctly.
* Subject has a history of fainting or vasovagal response.
* Subject has a history of sensitivity to local anesthesia
* Subject has a diagnosis of Raynaud's disease
* Subject has claustrophobia
* Subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
* Subject is pregnant, lactating or trying to get pregnant.
* Subject is unable or unwilling to provide informed consent or is unable or unwilling to comply with study procedures.
* Subject has any other condition, which in the opinion of the investigators would make them unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This was a prospective study with 12 healthy volunteers who met all the inclusion criteria and none of the exclusion criteria. Dormotech provided the investigational SpO2 sensors to conduct the evaluation with existing equipment at the site
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Measurement of arterial HbO2 saturations from 100% down to 70% | day 1
  At the start of each testing cycle, one blood sample was taken while breathing room air.
  Subjects then breathed through a partial rebreathing circuit with a nose clip, a mixture of nitrogen, air and carbon dioxide to reach six different stable levels (plateaus) of oxyhemoglobin saturation between 70-100%.

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Stratmann, MD PhD, Principal Investigator — Vital Signs Research Group, San Francisco, CA.
Locations (1):
- Vital Signs Research Group, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No